CLINICAL TRIAL: NCT01039051
Title: Randomized Controlled Trials of Diet and Lifestyle Intervention to Promote Chinese Postpartum Women's Health
Brief Title: Diet and Lifestyle Intervention Study in Postpartum Women in China
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Qingdao University (Other); Southern Medical University, China (Other); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Liegang Liu, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2008BA158B07
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Puerperal Infection; Fever; Constipation; Hemorrhoids; Anal Fissure; Breast Disease; Oral Ulcers; Anemia
MeSH Terms: conditions — Puerperal Infection; Fever; Constipation; Hemorrhoids; Fissure in Ano; Breast Diseases; Oral Ulcer; Anemia | interventions — Diet; Multicenter Studies as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diet and Lifestyle counseling (Experimental): increasing consumption of vegetables and fruits; maintaining energy balance through reducing excessive energy from meat, eggs and brown sugar and increasing energy expenditure from appropriate physical activity, such as doing maternal keep-fit exercises.
  Interventions: Behavioral: Diet and Lifestyle Intervention in Chinese Postpartum Women

INTERVENTIONS:
Behavioral: Diet and Lifestyle Intervention in Chinese Postpartum Women — For individual postpartum woman, we will set antepartum participatory training courses, provide specially prepared brochures and supporting VCD, set up a specialized counseling hotline and give individual bedside guidance after birth. For their family members, we will invite every postpartum woman's husband and mother to take part in workshops or seminars, making them know some basic knowledge of postpartum care, and persuading them to promote adoption of the diet and lifestyle we advocated by the postpartum woman. For community environment, we will put up posters about basic knowledge of postpartum care in the community bulletin boards for general population educating and mobilize community leaders and heads from and maternal and child health centers for maximum support.
  Other Names: Multicenter trial for Postpartum practice

SUMMARY:
Previous studies have shown "Doing the month", a traditional practice for postpartum women in China and other Asian countries, may be associated with higher prevalence of postpartum problems. The current multicenter randomized controlled trial (RCT) aims to evaluate outcomes of diet and lifestyle interventions in Chinese postpartum women.

DETAILED DESCRIPTION:
The current multicenter RCT will be conducted in three representative areas in China, Shandong province, Hubei province and Guangdong province, which locate in northern, central and southern parts of China, respectively. Women who attend routine pregnancy diagnosis in hospitals or maternal healthcare centers will be invited to take part in this study. At least 800 women who meet our eligibility criteria will be recruited and randomly assigned to the intervention group (n>=400) and the control group (n>=400). A three-dimension comprehensive intervention strategy, which incorporates intervention measures simultaneously to individual postpartum woman, their family members and community environment, will be utilized to maximize the effectiveness of intervention. Regular visiting and follow-up will be done in both group; nutrition and health-related measurements will be assessed both before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* at their third trimester
* had at least three routine examinations at these antenatal clinics

Exclusion Criteria:

* <20 or >40 years old

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1600 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the knowledge and belief about postpartum practice among the women | December 2009

SECONDARY OUTCOMES:
Changes in the nutritional status, postpartum recovery and health status | June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Liegang Liu, PhD, Study Chair — Huazhong University of Science and Technology
Locations (3):
- China (3):
  - Southern Medical University, Guangzhou, Guangdong
  - Huazhong University of Science and Technology, Wuhan, Hubei
  - Qingdao University, Qingdao, Shandong

REFERENCES:
- [Derived] Bao W, Ma A, Mao L, Lai J, Xiao M, Sun G, Ouyang Y, Wu S, Yang W, Wang N, Zhao Y, Fu J, Liu L. Diet and lifestyle interventions in postpartum women in China: study design and rationale of a multicenter randomized controlled trial. BMC Public Health. 2010 Feb 27;10:103. doi: 10.1186/1471-2458-10-103. PMID 20187965